CLINICAL TRIAL: NCT07344402
Title: A Prospective, Randomized, Controlled Trial Investigating Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) Intervention Strategies and Neurophysiological Mechanisms in Patients With Refractory Constipation
Brief Title: Optimization of taVNS Intervention Strategies for Refractory Constipation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Zhifeng Zhao, PhD, Principal Investigator, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XJLL-KY-20252521-2
Record Dates: First submitted 2025-12-23; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Refractory Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- taVNS (Experimental): Participants will receive active transcutaneous auricular vagus nerve stimulation (taVNS) delivered to the left cymba conchae using the study device. Stimulation will be administered twice daily for 20 consecutive days, with two 30-minute sessions per day separated by approximately 12 hours. Stimulation parameters will be 30 Hz with a 200 μs pulse width (single pulse width 200 μs).
  Interventions: Device: transcutaneous auricular vagus nerve stimulation
- Sham-tACS (Sham Comparator): Participants will receive a sham taVNS procedure designed to mimic active stimulation while not providing effective vagal nerve stimulation. Sham sessions will follow the same schedule and duration as the active arm: twice daily for 20 consecutive days, with two 30-minute sessions per day separated by approximately 12 hours. The sham condition will use an identical-appearing device and procedures to maintain blinding.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: transcutaneous auricular vagus nerve stimulation — Participants will receive active transcutaneous auricular vagus nerve stimulation (taVNS) delivered to the left cymba conchae using the study device. Stimulation will be administered twice daily for 20 consecutive days, with two 30-minute sessions per day separated by approximately 12 hours. Stimulation parameters will be 30 Hz with a 200 μs pulse width (single pulse width 200 μs).
  Arms: taVNS
Device: Placebo — Participants will receive a sham taVNS procedure designed to mimic active stimulation while not providing effective vagal nerve stimulation. Sham sessions will follow the same schedule and duration as the active arm: twice daily for 20 consecutive days, with two 30-minute sessions per day separated by approximately 12 hours. The sham condition will use an identical-appearing device and procedures to maintain blinding.
  Arms: Sham-tACS

SUMMARY:
The goal of this clinical trial is to learn whether transcutaneous auricular vagus nerve stimulation (taVNS) works to treat refractory constipation in adults. It will also learn about the safety and tolerability of taVNS. The main questions it aims to answer are:

Does taVNS improve constipation symptoms, as measured by the change in complete spontaneous bowel movements per week (ΔCSBMs/week) from baseline to post-treatment? What medical problems or side effects do participants have when receiving taVNS? Does taVNS reduce the need for rescue laxatives? Researchers will compare active taVNS to sham taVNS to see if taVNS works to treat refractory constipation.

Participants will:

Be randomly assigned (double-blind) to receive active taVNS or sham taVNS for 20 days Receive stimulation twice daily, 30 minutes per session, with a 12-hour interval between sessions Receive stimulation at 30 Hz with 200 μs pulse width, delivered to the left cymba conchae Keep a daily diary of bowel habits and symptoms, including CSBMs, and rescue laxative use (bowel movements occurring within 24 hours after rescue laxative use will not be counted as CSBMs)

ELIGIBILITY:
Inclusion Criteria (Revised) Diagnosis of Functional Constipation (FC): Meets Rome IV criteria for functional constipation.

Low CSBM frequency during screening: During the 2-week screening/run-in period, has ≤2 complete spontaneous bowel movements (CSBMs) per week, based on daily diary.

Inadequate response to prior therapy: History of ≥3 months of prior constipation treatment (e.g., laxatives and/or prokinetic agents) with inadequate response (persistent constipation symptoms and/or persistently low CSBM frequency) as documented by medical history and/or records.

Age: 18 to 80 years. Ability to comply: Able and willing to comply with study procedures (including stimulation sessions and diary completion).

No concurrent clinical trial participation: Not participating in another interventional clinical trial during the study period.

Informed consent: Provides written informed consent. Exclusion Criteria (Revised) Organic/secondary causes of constipation: Evidence or history of gastrointestinal organic disease (e.g., inflammatory bowel disease, colorectal tumor, congenital megacolon) or other conditions likely to cause secondary constipation, including endocrine/metabolic disorders (e.g., uncontrolled hypothyroidism, uncontrolled diabetes) or neurological disorders (e.g., Parkinson's disease, spinal cord disorders).

Medications causing constipation (unless stable): Current use of medications known to cause constipation (e.g., opioids, anticholinergics) that cannot be discontinued or kept stable during the study, in the investigator's judgment.

Opioid use disorder or chronic opioid use: History of substance abuse or chronic opioid use that may affect bowel function.

Severe psychiatric conditions or safety risk: Current severe psychiatric disorder requiring urgent intervention, or risk of self-harm/suicide as assessed by a qualified clinician.

Contraindications to taVNS or ear stimulation: Significant ear disease or skin lesions/infection at the stimulation site, or other contraindications to the study device/procedure.

Implanted electronic medical devices: Presence of implanted electrical devices (e.g., pacemaker, implantable cardioverter-defibrillator) or other conditions where electrical stimulation is contraindicated.

Pregnancy or lactation: Pregnant or breastfeeding women. Serious comorbidities that may interfere: Severe or unstable medical conditions that could interfere with participation or outcome assessment (e.g., significant cardiovascular disease/arrhythmia, coagulation disorders or regular anticoagulant therapy, severe hepatic/renal impairment, organ failure).

Cognitive/communication impairment: Cognitive impairment, aphasia, or other conditions preventing valid consent or reliable diary completion.

Investigator discretion: Any condition that, in the investigator's opinion, makes the participant unsuitable for the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
Predictive Value of Baseline EEG for Treatment Response (Area Under the Curve) | Baseline EEG predicting clinical outcome at Day 20
  The ability of baseline EEG spectral power (specifically alpha band power) to classify patients as Responders vs. Non-Responders. Responders are defined as patients with an increase of ≥1 CSBM/week. The performance will be assessed using Receiver Operating Characteristic (ROC) analysis.

SECONDARY OUTCOMES:
Change from baseline in weekly frequency of spontaneous bowel movements (SBM) | Baseline and end of treatment (Day 20)
Change in Complete Spontaneous Bowel Movements per Week (ΔCSBMs/week) | Baseline to end of treatment (Day 20)
  Primary efficacy outcome is the change in weekly complete spontaneous bowel movements (CSBMs) from baseline to end of treatment. A CSBM is defined as a spontaneous bowel movement accompanied by a sensation of complete evacuation. Weekly CSBMs will be derived from daily bowel diaries. Bowel movements occurring within 24 hours after use of rescue laxatives will not be counted as CSBMs.
Proportion of participants using polyethylene glycol (PEG) as rescue medication | Baseline and end of treatment (Day 20)
Change from baseline in Patient Health Questionnaire-9 (PHQ-9) score | Baseline and Day 20
Change from baseline in Generalized Anxiety Disorder-7 (GAD-7) score | Baseline and end of treatment (Day 20)
Change from baseline in Patient Health Questionnaire-15 (PHQ-15) somatic symptom score | Baseline and end of treatment (Day 20)

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi'an, China

IPD SHARING:
Plan to Share IPD: Yes
Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: For more information or to submit a request, please contact zhaozhifeng@outlook.com.